CLINICAL TRIAL: NCT05032430
Title: Reducing Maternal Stress to Improve Obesity-related Parenting Practices
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Virginia Commonwealth University (Other); George Washington University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Elizabeth Cotter, Assistant Professor, American University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-220-317; K23AT011049 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-09-02 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calma, Conversa, y Cría (CCC) (Experimental): Mindfulness-based parental stress reduction intervention
  Interventions: Behavioral: CCC
- Enhanced Usual Care (Active Comparator): Comparator group designed to influence health and well-being that does not include mindfulness as an active ingredient.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: CCC — A mix of mindfulness-based stress reduction, mindful eating, and mindful parenting strategies.
  Arms: Calma, Conversa, y Cría (CCC)
Behavioral: Enhanced Usual Care — Consists of strategies meant to enhance health and well-being (e.g., health education, strategies to get more physical activity) but does not include mindfulness as an active ingredient.
  Arms: Enhanced Usual Care

SUMMARY:
Maternal stress is associated with children's risk for obesity controlling for socioeconomic status. The association between maternal stress and child obesity is particularly strong in Latinx families, whose children also have the highest rates of obesity in the United States. A mindful parenting program might reduce Latina mothers' psychological stress and lead to improved parenting practices and ability to create a healthier environment. The primary objective of the proposed research is to evaluate the feasibility and acceptability of a culturally-relevant intervention that integrates mindfulness-based stress reduction and mindful parenting in Latina mothers. The investigators will conduct a randomized clinical trial comparing the Calma, Conversa, y Cría (CCC) intervention to an active control condition in 50 Latina mothers of elementary-school age children. Participant satisfaction rates and qualitative interviews will provide evidence of the program's acceptability. Feasibility will be determined by examining recruitment rates, retention rates, and treatment fidelity. Completion of this project will inform the development of a full-scale efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years
* identify as female
* identify as Hispanic or Latina
* have a child between the ages of 3 and 11 years who primarily resides with them
* able to understand basic instructions in either Spanish or English

Exclusion Criteria:

* pregnant or planning on becoming pregnant in the near future
* actively dependent on a substance
* have untreated psychosis, PTSD, or social anxiety that would impair their ability to function in a group setting
* child has an obesity-associated genetic syndrome
* child has a pervasive developmental disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 115 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-01-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with Intervention Assessed by the Client Satisfaction Questionnaire | Immediately after the intervention
  Parents will be asked to complete a brief, 8-item, widely used measure of satisfaction with health-related services, available in Spanish and English. Scores range from 8 to 32, with higher values indicating higher satisfaction.
Participant Retention | At the beginning of each of the 6 weekly intervention sessions
  Research staff will take attendance during each intervention session.

SECONDARY OUTCOMES:
Change in the Five Facet Mindfulness Questionnaire | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  The Five Facet Mindfulness Questionnaire (Spanish version) is a 39-item self-report measure of five facets of mindfulness: observing, describing, acting with awareness, non-judgment, and non-reactivity. Scores range from 39 to 190 with higher scores suggesting greater mindfulness.
Change in the Perceived Stress Scale | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  The Perceived Stress Scale is a 10-item, widely used self-report measure of perceptions of psychological stress. Scores range from 0 to 40 with higher scores indicating greater perceived stress.
Change in the Child Feeding Questionnaire | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  The Child Feeding Questionnaire is a 31-item self-report questionnaire that assesses parents' beliefs, attitudes, and approaches toward feeding their children. Scores range from 31 to 155 with higher scores representing greater use of controlling feeding practices.
Change in the Frequency of Family Eating and Exercise Behaviors Questionnaire | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  28 items used in previous work by Neumark-Sztainer et al. will be used to assess eating and weight-related habits of families. Items assess: frequency of family meals, fast food consumption, and watching TV during meals; availability of fruits and vegetables and sugar sweetened beverages; and parents' encouragement of healthy food consumption and physical activity.
Change in height in meters | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Height will be measured to the nearest 0.1cm using a precision stadiometer.
Change in weight in kilograms | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Weight will be measured to the nearest 0.1kg using a digital scale.

OTHER OUTCOMES:
Change in Child Daily Kilocalories via 3-Day Food Record | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Participants will be trained to complete a 3-day food record (using a detailed food record form) to track dietary intake for 2 weekdays and 1 weekend day in the week prior to their assessment. Diet will be analyzed via Nutrition Data System Software (NDSR). Average kilocalories per day will be the primary dietary outcome.
Change in Child Frequency of Physical Activity as Assessed by the Physical Activity Recall Screen | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Children's frequency of physical activity will be assessed using the Physical Activity Recall. This interview measure asks respondents to report the amount of time they spent in moderate and vigorous activities during the previous 7 days.
Change in Child Quality of Life as Assessed by the Pediatric Health-Related Quality of Life Questionnaire | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  The Pediatric Quality of Life Questionnaire is a 23-item measure of perceptions of how health affects daily life in 4 areas: physical, emotional, social, and school. Scores range from 0 - 100, with higher scores indicating greater quality of life.
Change in Child Weight in Kilograms | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Weight will be measured to the nearest 0.1kg using a digital scale.
Change in Child Height in Meters | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Height will be measured to the nearest 0.1cm using a precision stadiometer.
Change in Accelerometry | Participants will complete this at three timepoints: baseline, immediately after the intervention, and 10-months from baseline
  Accelerometers (Actigraph GT3X) will be worn for 1 week by children for each assessment period to assess physical activity objectively.

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided